CLINICAL TRIAL: NCT00610844
Title: Evaluation of Effectiveness of Preoperative Percutaneous Radiofrequency Ablation of Primary and Secondary Lung Tumors
Brief Title: Preoperative Percutaneous Radiofrequency Ablation of Primary and Secondary Lung Tumors
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Hospital Tuebingen (Other)
Responsible Party: Philippe L. Pereira, MD, Department of Diagnostic Radilogy
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LungRFA_V1
Record Dates: First submitted 2008-01-28; First posted 2008-02-08 (Estimated); Last update posted 2008-02-20 (Estimated); Status verified 2007-11

CONDITIONS: Lung Cancer; Lung Metastasis
Keywords: lung cancer; lung metastasis; radiofrequency ablation
MeSH Terms: conditions — Lung Neoplasms

ARMS (1):
- 1 (Experimental): pulmonary radiofrequency ablation
  Interventions: Procedure: pulmonary radiofrequency ablation

INTERVENTIONS:
Procedure: pulmonary radiofrequency ablation — CT-guided pulmonary radiofrequency ablation

SUMMARY:
The purpose of the study is to evaluate the effectiveness of radiofrequency ablation by pathological correlation and to characterize the tissue response after treatment of primary and secondary pulmonary tumors.

DETAILED DESCRIPTION:
Thermal ablation therapy is an increasingly performed technique in the local tumor treatment. Among these techniques, image-guided radiofrequency (RF) ablation attained widespread consideration in the therapy of liver tumors and osteoid osteoma. Promising results of hepatic RF ablation raised expectations to utilize the advantages of image-guided ablation therapy for the treatment of pulmonary malignancies. The purpose of the study is to evaluate the effectiveness of radiofrequency ablation by pathological correlation and to characterize the tissue response after treatment of primary and secondary pulmonary tumors. Computed tomography-guided RF ablation is performed in local or general anesthesia, followed by surgical resection three days later. An analysis of complete RF ablation and a characterization of tissue response is performed by hematoxylin and eosin staining, immunostaining, and electron microscopy. Adverse effects and complications are recorded.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent for radiofrequency ablation and surgery
* Maximum of 3 lung tumors
* Maximum tumor size 5 cm
* Must be able to receive standard surgery

Exclusion Criteria:

* Pathological coagulation tests
* Pregnant or breast feeding
* Maximum tumor size more than 5 cm
* Bilateral secondary lung cancer with more than 3 tumors
* Inoperable patient

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2004-04; Primary Completion 2006-05 (Actual)

PRIMARY OUTCOMES:
rate of incomplete treated tumors | 3 days

SECONDARY OUTCOMES:
pathologic tissue changes, rate of major and minor complications | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Philippe L Pereira, MD, Principal Investigator — Department of Diagnostic Radiology, University of Tübingen; Hermann Aebert, MD, Principal Investigator — Department of thoracic surgery, University of Tübingen
Locations (1):
- Department of Diagnostic Radiology, Tübingen, Baden-Wurttemberg, Germany